CLINICAL TRIAL: NCT06314282
Title: INTERSTELLAR - Multi-National, Observational, Prospective, Post-Launch, Effectiveness Study Among SLE Patients Receiving Anifrolumab in Routine Clinical Practice
Brief Title: INTERSTELLAR - International Study Evaluating Lupus Outcomes After Anifrolumab Real World Use
Acronym: INTERSTELLAR
Status: Recruiting | Type: Observational
Sponsor: AstraZeneca (Industry)
Responsible Party: Sponsor
Other Study IDs: D3461R00072
Record Dates: First submitted 2024-03-11; First posted 2024-03-18 (Actual); Last update posted 2026-01-15 (Actual); Status verified 2026-01

CONDITIONS: Systemic Lupus Erythematosus (SLE)
Keywords: SLE; Systemic lupus erythematosus; autoimmune disease; Lupus; Anifrolumab
MeSH Terms: conditions — Lupus Erythematosus, Systemic; Autoimmune Diseases

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
INTERSTELLAR study will generate critical prospective real-world evidence on the benefits of adding Anifrolumab to standard of care treatment for SLE in routine clinical practice, to inform physicians, payers and patients. The study will use clinical assessments that are relevant for SLE-treating physicians in routine clinical practice, as well as introduce a specific measure for skin manifestations to affirm the potency of anifrolumab in treating SLE-related skin manifestations. The study will use standardized objectives, inclusion/exclusion criteria and outcome measures across all countries participating in this study including GCC (Qatar, KSA), Mexico, CAMCAR (Costa Rica, Panama, Dominican Republic), Colombia, Argentina, Taiwan, and Egypt, and any other countries that may be included in the study, in order to facilitate a comparison and analysis across all countries included in this study.

DETAILED DESCRIPTION:
INTERSTELLAR is a multi-country, single-arm, observational, cohort study, with 1 year retrospective baseline data and 1 year of prospective follow-up. The study will be initiated on a country-by-country basis following the commercial launch of anifrolumab. The enrolment period is anticipated to be 12 months per country. In general, patients will enter the study between the first anifrolumab prescription and infusion (index), with follow-up until death, loss to follow-up, patient discontinuing the study, or end of study period (whichever occurs first). Relevant clinical and patient reported outcome (PRO) data collection for the entire follow up will continue for patients who have discontinued anifrolumab during the study, unless the patients have withdrawn their consent for participation in the study

ELIGIBILITY:
Inclusion Criteria:

1. Aged 18 years or older at study enrolment.
2. Fulfilled the 2019 EULAR/ACR criteria1 for SLE at the time of study entry.
3. Prescribed anifrolumab for their SLE treatment for the first time, according to approved country-specific label.
4. It is important to note that a physician decision to prescribe anifrolumab will need to occur prior to any study-related discussion.
5. In countries where prescription reimbursements are authorized on a case-by-case basis, authorization (ie, patient access to treatment) will be required for study entry.
6. Provided informed consent to participate in the study.
7. Willing and able to participate in all required study evaluations and procedures.

Exclusion Criteria:

1. Currently participating in an anifrolumab early access/compassionate use program or an interventional clinical trial with an investigational product.
2. Previous exposure to anifrolumab as part of a clinical trial or early access program.
3. Documented diagnosis of severe or rapidly progressive Class III or IV glomerulonephritis requiring induction therapy (mycophenolate mofetil [MMF]/cyclophosphamide [CYC] + high dose steroids), isolated Class V lupus nephritis, or active severe or unstable neuropsychiatric lupus.
4. Any other condition which the investigator deems to limit a patient's ability to understand the informed consent or complete the PROs.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: 10 to 50 patients will be enrolled per country from academic, community and hospital outpatient settings, to maximize the representation of the study population. This will result in approximately 180-200 patients in total allowing for sufficient precision when analysing the total cohort and to explore subgroups of interest.
Sampling Method: Non-Probability Sample
Enrollment: 200 (Estimated)
Dates: Start 2024-10-22 (Actual); Primary Completion 2027-03-31 (Estimated); Study Completion 2027-03-31 (Estimated)

PRIMARY OUTCOMES:
PGA | Baseline (pre-infusion) Month 1, Month 3, Month 6, Month 12
  Physician's overall assessment of disease activity on a visual analog scale ranging from 0 (no activity) to 3 (severe activity).
SLEDAI-2K | Baseline (pre-infusion) Month 1, Month 3, Month 6, Month 12
  24 lupus-related (weighted) items to assess disease activity, rated as 'present' or 'absent' and attributed to active lupus. Scored on a scale from 0 to 105, with 0 being inactive disease.
CLASI | Baseline (pre-infusion) Month 1, Month 3, Month 6, Month 12
  Skin activity and damage assessment completed by physician by scoring each specific area as indicated on the form. The higher the score, the worse the activity/damage.
FACIT-Fatigue | Baseline (pre-infusion) Month 1, Month 3, Month 6, Month 12
  A 13-item questionnaire to assess the impact of fatigue on a 5-point verbal rating scale. Scores range from 0 to 52; a higher score indicates les fatigue
LupusQoL | Baseline (pre-infusion) Month 3, Month 6, Month 12
  A 34-item questionnaire on a verbal rating scale covering several domains, including daily activities, pain, fatigue and sleep in relation to lupus symptoms.
EQ-5D-5L | Baseline (pre-infusion) Month 3, Month 6, Month 12
  5-item questionnaire measuring 5 dimensions of general health status on a verbal rating, and a single visual analog scale about overall perceived health today

CONTACTS AND LOCATIONS:
Locations (14):
- Argentina (2):
  - Research Site, Buenos Aires
  - Research Site, Córdoba
- China (3):
  - Research Site, Guangzhou
  - Research Site, Shenzhen
  - Research Site, Zhongshan
- Research Site, Muscat, Oman
- Research Site, Doha, Qatar
- Saudi Arabia (3):
  - Research Site, Abhā
  - Research Site, Jeddah
  - Research Site, Riyadh
- Taiwan (4):
  - Research Site, Kaosiung
  - Research Site, New Taipei City
  - Research Site, Taichung
  - Research Site, Taipei

IPD SHARING:
Plan to Share IPD: Yes
Qualified researchers can request access to anonymized individual patient-level data from AstraZeneca group of companies sponsored clinical trials via the request portal.
  All request will be evaluated as per the AZ disclosure commitment:
  https://astrazenecagrouptrials.pharmacm.com/ST/Submission/Disclosure Yes, indicates that AZ are accepting requests for IPD, but this does not mean all requests will be shared.
Time Frame: AstraZeneca will meet or exceed data availability as per the commitments made to the EFPIA Pharma Data Sharing Principles. For details of our timelines, please rerefer to our disclosure commitment at https://astrazenecagrouptrials.pharmacm.com/ST/Submission/Disclosure.
Access Criteria: When a request has been approved AstraZeneca will provide access to the deidentified individual patient-level data in an approved sponsored tool . Signed Data Sharing Agreement (non-negotiable contract for data accessors) must be in place before accessing requested information. Additionally, all users will need to accept the terms and conditions of the SAS MSE to gain access. For additional details, please review the Disclosure Statements at https://astrazenecagrouptrials.pharmacm.com/ST/Submission/Disclosure.
URL: https://astrazenecagroup-dt.pharmacm.com/DT/Home